CLINICAL TRIAL: NCT01514773
Title: Patient and Physician Knowledge and Attitudes Toward Defibrillator Therapy Survey Study
Brief Title: Patient and Physician Survey Determinants of Appropriate ICD Utilization
Status: Completed | Type: Observational
Sponsor: Todd M Koelling, MD (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Todd M Koelling, MD, Associate Professor, Director Heart Failure Program, University of Michigan
Organization: University of Michigan (Other)
Other Study IDs: HUM00050147
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure, Systolic
Keywords: left ventricular systolic dysfunction; implantable cardioverter defibrillator; systolic heart failure; congestive heart failure; Ischemic cardiomyopathy; Nonischemic cardiomyopathy; ICD; ICD utilization; ICD implantation; defibrillator; defibrillator therapy; sudden cardiac death
MeSH Terms: conditions — Heart Failure, Systolic; Ventricular Dysfunction, Left; Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICD placement: Those subjects who have an ICD.
- No ICD placement: Those subjects who have not had an ICD placed.

SUMMARY:
To better understand the reasons for underutilization of defibrillator therapy in selected populations, the investigators propose a study to assess heart failure patient knowledge and attitudes toward device therapy. By carefully studying populations of patients with systolic heart failure, the investigators aim to identify the underlying reasons for implantable cardioverter defibrillators (ICD) non-utilization in patients with symptomatic systolic heart failure.

DETAILED DESCRIPTION:
Several multi-center randomized trials have demonstrated the benefit of implantable cardioverter defibrillators (ICDs) for the primary prevention of sudden cardiac death among patients with ischemic and nonischemic cardiomyopathy. Guideline documents for the treatment of heart failure have recommended defibrillator placement for patients with symptomatic heart failure and left ventricular ejection fraction (LVEF) ≤ 35%. Despite these recommendations, observational studies have documented low ICD utilization among patients with heart failure. Recent studies have demonstrated patient specific characteristics that are associated with low ICD utilization (advanced age, female gender, black race, heart failure etiology, uninsured patients and patients cared for by general practitioners). Whether patient knowledge or attitudes regarding defibrillator therapy influence the rate of defibrillator placement is unknown. By carefully surveying populations of patients with systolic heart failure, we aim to further the understanding of the patient factors that determine why an ICD may or may not be used in the appropriate clinical setting. Additionally, 150 physicians will be enrolled into the study for the purpose of measuring attitudes and beliefs regarding defibrillator treatment for the physicians providing care to the patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Left ventricular ejection fraction ≤ 35%
* Previous diagnosis of heart failure with current NYHA Class II-III symptoms
* Established UMHS patient with at least two outpatient visits in the past two years to either Primary Care or Cardiology, OR, at least one inpatient admission in the past two years along with at least one outpatient visit within the past 13 months to Primary Care or Cardiology

Exclusion Criteria:

* Patients having undergone heart transplantation
* Patients having undergone placement of a left ventricular assist device
* Patients with congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of Michigan Health System Ambulatory Heart Failure Registry
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2013-08-30 (Actual); Study Completion 2013-08-30 (Actual)

PRIMARY OUTCOMES:
Patient Determinants of Appropriate ICD Utilization | 1 year
  Specifically, we will assess patients for knowledge deficits regarding the clinical effects of ICD therapy. We will assess patients for their opinions regarding their risk of death, and whether they are willing to trade time to avoid discomfort of their illness or ICD shocks. We will ask patients about their thoughts about financial concerns regarding ICD therapy and their trust in technology, their physician and the medical system. We will also ask patients about their opinions regarding cosmetic issues created by ICD placement.

SECONDARY OUTCOMES:
Physician Determinants of Appropriate ICD Utilization | 1 year
  Measure physician knowledge and attitudes regarding defibrillator therapy for the physicians providing care to the patients in the study and assess the relationship between these measures and appropriate defibrillator utilization. We will assess physicians understanding of ICD clinical effects, costs, and risks of complications.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Koelling, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States